CLINICAL TRIAL: NCT00873054
Title: Percutaneous Nephrolithotomy Versus Extracorporeal Shock Wave Lithotripsy
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Samuel Deem, DO, Principal Investigator, CAMC Health System
Other Study IDs: 08-08-2078
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 ESWL: In this procedure,scope will be placed inside bladder and a plastic tube (stent) will be left to drain the kidney on the affected side in a routine manner. Next the patient will be transferred to a separate room and sound waves will be aimed at the center of the stone until the stone is broken into pieces.
- 2 PCNL: In this procedure,scope will be placed inside bladder and a plastic tube (stent) will be left to drain the kidney on the affected side in a routine manner. Next, a small (1cm) cut will be made in the back and a tube will be placed into the kidney. Through this tube a small camera will be placed inside the kidney and break the stone into many pieces and remove them through the same tube. All fragments that can be seen will be removed. A different plastic tube (drain) will be placed through the cut and into the kidney and left in place for 5-7 days.

SUMMARY:
The investigators main hypothesis is that the stone free rate will be much higher (95%) in patients treated with PCNL than patients treated with ESWL where stone free rate is (60%) to determine which treatment is safe and prevent less stone recurrence.

DETAILED DESCRIPTION:
Extracorporeal shock wave lithotripsy is preferred for small stones less than 10 mm in size. Percutaneous nephrolithotomy is the standard therapy used for large kidney stones greater than 20 millimeters or stones in the lower kidney. For moderate sized kidney stone (10-20 mm),currently the options for treatment include both methods. However, no studies have proven that one procedure is better than the other. So, we will compare both the procedures for breaking the kidney stone. Our main outcome measures will be the stone-free status after the procedure. Other outcome measures are assessment of morbidity associated with use of the procedures i.e. any minor or major complications within 3 months of initial treatment. Patient will be assessed for infection at post-operative office visits to include a basic urinalysis only if they have systemic indicators of infection (fever, dysuria, frequency, etc.). Pain will be monitored with the scale of 0-10 points. Also we will review of stone density on Computerized Tomography (CT) scans and the effect this has on success of both procedures. We hope with PCNL stone-free rates will be minimum with minimal morbidity and ultimately improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex with age greater than 18 years to 90 years
* Stone burden between 10 and 20 mm diagnosed by CT scan
* Patient must be agreeable to randomization between shock wave lithotripsy and percutaneous stone removal

Exclusion Criteria:

* Patients with bleeding diathesis or taking anti-platelet or anti-coagulant medication
* Patients who are pregnant based on routine pre-operative pregnancy testing
* Patients with skin to stone size greater than 12 cm (measured routinely on CT scan)
* Patients with either Horseshoe kidney, transplant kidney or a solitary kidney
* Patients with ureteral calculi
* Patients with stone size of < 10 mm and > 20 mm
* Ureteropelvic junction obstruction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community patients who present to Charleston Area Medical Center (CAMC) or the private urology clinics of Drs. Tierney, Martinez or Davalos with kidney stones between 10 and 20 mm in size would be screened based on inclusion criteria for possible enrollment in the study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the stone-free status after Extracorporeal Shock Wave Lithotripsy (ESWL) and Percutaneous Nephrolithotomy (PCNL) for kidney stones 10-20 mm in size. | Within 3 months of enrollment

SECONDARY OUTCOMES:
A secondary objective is to assess the morbidity associated with use of the procedures i.e. any minor or major complications within 3 months of initial treatment. | Within 3 months of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Julio G. Davalos, MD, Principal Investigator — CAMC Medical Staff - with admitting privileges; Frederick Martinez, M.D., Principal Investigator — CAMC Medical Staff - with admitting privileges
Locations (1):
- Urology Center of Charleston, Charleston, West Virginia, United States

REFERENCES:
- [Derived] Setthawong V, Srisubat A, Potisat S, Lojanapiwat B, Pattanittum P. Extracorporeal shock wave lithotripsy (ESWL) versus percutaneous nephrolithotomy (PCNL) or retrograde intrarenal surgery (RIRS) for kidney stones. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007044. doi: 10.1002/14651858.CD007044.pub4. PMID 37526261